CLINICAL TRIAL: NCT05546541
Title: Nutrition as a Risk Factor and Predictor of the Outcome of Orthobiological Treatments for Knee Osteoarthritis
Brief Title: Epidemiology and Nutrition
Acronym: Nutririsk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Nutririsk
Record Dates: First submitted 2021-12-28; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Diseases; Osteoarthritis, Knee; Nutrition, Healthy
MeSH Terms: conditions — Musculoskeletal Diseases; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- subjects normal weight undergo to PRP treatment: subjects with body mass index (BMI) considered normal weight (≥18.5 and ≤25) undergo to Platelet-Rich Plasma (PRP) treatment.
- subjects overweight undergo to PRP treatment: subjects with BMI values that exceed the normal weight range (BMI>25) undergo to PRP treatment.
- subjects with normal weight undergo to microfragmented adipose tissue treatment: subjects with BMI within the considered normal weight range (≥18.5 e ≤25) and undergo to microfragmented adipose tissue treatment.
- subjects overweight undergo to microfragmented adipose tissue treatment: subjects with BMI values that exceed the normal weight range undergo to microfragmented adipose tissue treatment. (BMI>25).

SUMMARY:
The general purpose of this study is to evaluate the relation between the nutritional status of patients, the features of the orthobiologics products used for patients' treatment and the clinical outcomes after one-step conservative regenerative treatment for knee osteoarthritis.

DETAILED DESCRIPTION:
The general purpose of this monocentric, observational with additional procedure (extra routine blood sampling, questionnaires and measurement of Nutritional status), prospective and non-controlled study is to evaluate the relation between the nutritional status of patients, the features of the orthobiologics products used for patients' treatment and the clinical outcomes after one-step conservative regenerative treatment (Platelete rich plasma and micro-fragmented adipose tissue injections) for knee osteoarthritis.The primary outcome of the study will be the identification of the proportion of responders and non-responders patients to the orthobiologic treatment (according to OMERACT-OARSI criteria) at 6-month follow-up. Another primary outcome will be the nutritional status identification of the same patients.

For these purposes the responder or non-responder patients will be identified based on the results of the Visual Analogue Scale (VAS) [the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100; a higher score indicates greater pain intensity no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)], Tegner-Lysholm Activity Scale and Knee Injury (Scores range from 0=worse disability to 100=less disability) and Osteoarthritis Outcome score (KOOS) (the score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems) according to the parameters established by Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) and Osteoarthritis Research Society International (OARSI) [they cannot be represented by a range of values]. The secondary outcomes of the study will be:

* the identification of the proportion of responders and non-responders patients to the orthobiologic treatment (according to OMERACT-OARSI criteria) at 2 and 12-month follow-up and of their related nutritional status;
* the characterization of the orthobiologic products used for the patient's treatment.

After the ethics committee approval, patients meeting the inclusion criteria undergoing conservative knee regenerative medicine treatments with orthobiologics and participating to the observational study "REGAIN" will be enrolled into the study. The PROMs will be completed by patients based on their clinical condition and on the specific treatment they will receive at the REGAIN Center. The aforementioned PROMs include but are not limited to:

- VAS, Tegner-Lysholm Activity Scale, KOOS. Patients will be asked to filled the PROMs at the time of the enrollment (before the treatment) and then at 2, 6 and 12 months after the treatment.

Blood and nutritional information will be collected only the day of the treatment to allow for evaluation of the possible association between patients' characteristics and treatment outcomes. Blood sampling will be performed to carry out the following laboratory analysis, in detail: complete blood count (cell number/dl), blood glucose (mg/dl), hemoglobin A1C (HbA1c) (mmol/mol), creatinine (mg/dl), Glutamic Oxaloacetic Transaminase (GOT) and Glutamic-Pyruvic Transaminase (GPT) (U/L), C reactive protein (mg/dl), triglycerides (mg/dl), total cholesterol(mg/dl), HDL(mg/dl).

In particular, for patients undergoing a Platelet Rich Plasma (PRP) treatment, a blood sample is already routinely harvested and therefore only an extra test tube will be added to test blood glucose (mg/dl), hemoglobin A1C (HbA1c) (mmol/mol), creatinine (mg/dl), GOT and GPT transaminases (U/L), C reactive protein (mg/dl), triglycerides (mg/dl), total cholesterol(mg/dl), HDL(mg/dl). For patients undergoing a treatment with microfragmented adipose tissue, an ad hoc blood collection will be carried out by filling two test tubes.

Nutritional information include anthropometric measurements, diet history and food consumption questionnaire (24h recall, "How much do i really eat?", Italian Mediterranea Index, anamnesi). Anthropometric measurements include weight (kg) and height (m), waist circumference (cm), arm circumference measurements (cm), biceps, triceps, subscapular and suprailiac folds measurement (mm) (plicometry) through the use of the skinfolder. It should be noted that the skinfolder is only one of the tools used to evaluate the patient's nutritional status, without diagnostic purposes and without the will to investigate anything about the device.

Concerning the orthobiologics characterization, PRP and microfragmented adipose tissue will undergo to different evaluations as per the observational study protocol "REGAIN".

In addition, for the purpose of this study, isolation and characterization of extracellular vesicles derived from PRP and micro fragmented adipose tissue will be performed, in order to deepen the orthobiologic characterization. The following techniques will be applied, where appropriate:

* Count and identification of cells from PRP and microfragmented adipose tissue (hemacytometer, nucleocounter, flow cytometry);
* Extracellular vesicle isolation, count and dimensional analysis (ultracentrifuge, Nanosights);
* Extracellular vesicle marker identification (flow cytometry).

These data will be analyzed for their possible association with nutritional status of the patient and clinical outcomes.

Regardless the specific protocol or investigation, the analysis will not include genomic DNA or diagnostic analysis. All samples (blood and tissues) will be analyzed at Istituto Ortopedico Galeazzi and destroyed at the end of the study. Total duration of this study is of 36 months after approval of Ethical Committee.

ELIGIBILITY:
Inclusion Criteria:

* males and females ≥18 and ≤ 65 years;
* presence of knee osteoarthritis;
* indication to regenerative medicine treatments PRP or microfragmented adipose treatment;
* participation to the observational study "REGAIN";
* patients with BMI ≥18.5;
* signature of Informed Consent for the study.

Exclusion Criteria:

* patients with BMI <18.5;
* patients who are not able to comply with the study schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by knee osteoarthritis undergoing conservative regenerative medicine procedures with autologous material at IRCCS Istituto Ortopedico Galeazzi and participating to the observational study "REGAIN" will be enrolled for this study:
  88 patients will be needed:
  1. 22 subjects with body mass index (BMI) considered normal weight (≥18.5 and ≤25) undergo to Platelet-Rich Plasma (PRP) treatment;
  2. 22 subjects with BMI>25 undergo to PRP treatment;
  3. 22 subjects with BMI ≥18.5 and ≤25 undergo to microfragmented adipose tissue treatment;
  4. 22 subjects with BMI >25 undergo to microfragmented adipose tissue treatment.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
6 months follow-up, responders and not responders | 6 months after treatment
  Identification of the proportion of responders and non-responders patients to the orthobiologic treatment (according to OMERACT-OARSI criteria) at 6-month follow-up.
Identification of the nutritional status of patients: Complete blood count | 10 minutes before the treatment
  Complete blood count (cell number/dl)
Identification of the nutritional status of patients: Blood glucose | 10 minutes before the treatment
  Blood glucose (mg/dl) measurement
Identification of the nutritional status of patients: blood Hemoglobin A1C (HbA1c) | 10 minutes before the treatment
  Hemoglobin A1C (HbA1c) (mmol/mol) measurement
Identification of the nutritional status of patients: blood creatinine | 10 minutes before the treatment
  Creatinine (mg/dl) measurement
Identification of the nutritional status of patients: blood Glutamic-Oxaloacetic Transaminase GOT (U/L) | 10 minutes before the treatment
  Glutamic-Oxaloacetic Transaminase GOT (U/L) measurement
Identification of the nutritional status of patients: blood Glutamate Pyruvate Transaminase GPT | 10 minutes before the treatment
  Glutamate Pyruvate Transaminase GPT (U/L) measurement
Identification of the nutritional status of patients: blood C reactive protein | 10 minutes before the treatment
  C reactive protein (mg/dl) measurement
Identification of the nutritional status of patients: blood Triglycerides | 10 minutes before the treatment
  Triglycerides (mg/dl) measurement
Identification of the nutritional status of patients: blood total cholesterol | 10 minutes before the treatment
  Total cholesterol (mg/dl) measurement
Identification of the nutritional status of patients: blood High Density Lipoprotein HDL | 10 minutes before the treatment
  High Density Lipoprotein HDL (mg/dl) measurement
Anthropometric measurement: weight | 10 minutes before the treatment
  weight (kg) measurement
Anthropometric measurement: height | 10 minutes before the treatment
  height (m) measurement
Anthropometric measurement: waist circumference | 10 minutes before the treatment
  waist circumference (cm) measurement
Anthropometric measurement: arm circumference measurements | 10 minutes before the treatment
  arm circumference measurements (cm)
Anthropometric measurement: biceps folds measurement | 10 minutes before the treatment
  biceps folds measurement (mm)
Anthropometric measurement: triceps folds measurement | 10 minutes before the treatment
  triceps folds measurement (mm)
Anthropometric measurement: subscapular folds measurement | 10 minutes before the treatment
  subscapular folds measurement (mm)
Anthropometric measurement: suprailiac folds measurement | 10 minutes before the treatment
  suprailiac folds measurement (mm)

SECONDARY OUTCOMES:
2 months follow-up, responders and not responders | 2 months after treatment
  The identification of the proportion of responders and non-responders patients to the orthobiologic treatment (according to OMERACT-OARSI criteria) at 2 months follow-up
12 months follow-up, responders and not responders | 12 months after treatment
  The identification of the proportion of responders and non-responders patients to the orthobiologic treatment (according to OMERACT-OARSI criteria) at 12 months follow-up
The characterization of the orthobiologic products. | 15 minutes after the treatment
  The characterization of the orthobiologic products used for the patient's treatment that include isolation and characterization of extracellular vesicles derived from PRP and micro fragmented adipose tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Galeazzi orthopaedic institute, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT05546541/Prot_000.pdf